CLINICAL TRIAL: NCT00156611
Title: ReoPro and Peripheral Arterial Intervention to Improve Clinical Outcome in Patients With Peripheral Arterial Disease - A Randomized Prospective Trial (RIO-Trial)
Brief Title: Rio Trial - ReoPro and Peripheral Arterial Intervention to Improve Clinical Outcome in Patients With Peripheral Arterial Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University of Bern (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R-1
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2006-09-12 (Estimated); Status verified 2006-09

CONDITIONS: Arterial Occlusive Diseases
Keywords: peripheral vascular disease; intervention; restenosis; Age above 18 years
MeSH Terms: conditions — Arterial Occlusive Diseases; Peripheral Vascular Diseases | interventions — Angioplasty, Balloon; Abciximab

INTERVENTIONS:
Procedure: Balloon Angioplasty
Drug: ReoPro

SUMMARY:
The Rio Study is a randomized, double blinded German- Swiss- Austria multi-centre trial on the efficacy and safety of ReoPro together with interventional recanalization of TASC D lesions in the SFA and popliteal artery.

DETAILED DESCRIPTION:
Purpose: The RIO trial is designed to test the efficacy of GP IIb/IIIa blockade on subacute reocclusions in patients with interventional recanalization of chronic occlusions in the superficial femoral and popliteal artery.

Methods: A total of 420 patients will be randomly assigned to ReoPro or placebo. Patients will be eligible for randomisation with occlusions longer than 5 cm. Doppler ultrasound follow-up will be at 30 days, and after 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of peripheral artery disease with superficial femoral or popliteal artery occlusion, which mandates PTA or stent administration as first treatment modality. The history of peripheral artery occlusion has to be at least 6 weeks, and the target vessel occlusion has to be more than 5 centimeters in length.
* Age between 18 and 90 years

Exclusion Criteria:

* Acute limb ischemia
* Subacute ischemia with requires thrombolysis as first treatment modality
* Active bleeding or known bleeding diathesis
* Known severe hepatic or renal disorder (liver cirrhosis, stage B, C or serum creatinine > 2.5 mg%)
* Hyperthyreosis
* Diabetes mellitus treated with metformin
* Known heparin induced thrombocytopenia (HIT, type 2)
* Female sex with childbearing potential
* Major surgery or trauma in past 6 weeks
* History of stroke within the previous 2 years, or any stroke with a residual neurological deficit, or other CNS abnormality (e.g., intracranial neoplasm, arteriovenous malformation, or aneurysm)
* Gastrointestinal or genitourinary bleeding of clinical significance within the previous 6 weeks
* Administration of oral anticoagulants within the previous 7 days unless prothrombin time is < 1.2 times control (or international normalized ratio [INR] <1.4), or ongoing treatment with oral anticoagulants
* History of bleeding diathesis of platelet count < 100,000/mm3
* Arteriovenous malformations or aneurysms
* Severe uncontrolled hypertension (treated sys. BP > 200 mm Hg, diast. BP > 100 mm Hg)
* Hypertensive or diabetic retinopathy
* Vasculitis
* Known autoimmune disorders
* Patient with aspirin intolerance
* Contraindication or known allergic reactions to abciximab or murine proteins
* Co-existent condition associated with a limited life expectancy (e.g., advanced cancer, end-stage congestive heart failure)
* Participation in another clinical research study involving the evaluation of another investigational drug or device within 7 days prior to enrollment
* Patient who has previously received a GP IIb/IIIa antagonist

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420
Dates: Start 2002-01; Study Completion 2009-12

PRIMARY OUTCOMES:
Prevention of subacute occlusions within 30 days

SECONDARY OUTCOMES:
Prevention of restenosis up to 3 years
Prevention of target lesion revascularization
Improvement of the clinical status
Change of ABI
Hospital days
all secondary outcomes at 30 days, 6 months, one year, and 3 years (telephone contact after 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, MD, Principal Investigator — University Hospital of Tuebingen; Iris Baumgartner, MD, Principal Investigator — University of Bern
Locations (1):
- University of Tuebingen, Tübingen, Germany